CLINICAL TRIAL: NCT07138300
Title: Combined Effect of Low Level Laser Therapy and Neural Mobilization on Lumber Disc Prolapse
Acronym: LLLT-NM-LDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, assistant professor , department of physical therapy for musculoskeletal disorders and its surgeries, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC\012\004894
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Low Level Laser Therapy
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Masking Description: the patient and the research assistant are blind about the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (B) (Experimental): 20 patients will receive low level laser therapy plus neural mobilization.
  * Mobilization will be through using slump sitting maneuver (Both techniques
    1. The slider neurodynamic mobilization technique:
       The patient moves actively and conversely from a position of neck and trunk flexion, knee flexion, and ankle plantar flexion, to a position of neck and trunk extension, knee extension and ankle dorsiflexion.
    2. The tension neurodynamic mobilization technique:
       The patient moves actively and conversely from a position of neck and trunk extension, knee flexion, and ankle plantar flexion, to a position of neck and trunk flexion, knee extension, and ankle dorsiflexion
  * Low level laser therapy : Twenty points were established for treatment, 12 over the lumbar spine, at the same Side of the radicular pain, from l2 to s1 vertebra, distance between these points is 2 cm. In the thigh, eight points were marked at equal distances from each other, four in the path of l5 root and four in the path of
  Interventions: Device: Low Level Laser Therapy by (Eme Physio, Lasermed 2200), GaAs laser, 1 cm2 beam area,7,000 Hz, 17 mW, 1 J/cm2, Pesaro, Italy); Procedure: neural mobilization
- control group (A) (Active Comparator): 20 will receive placebo laser therapy plus neural mobilization. Mobilization will be through using slump sitting maneuver (Both techniques slider and tensioner.
  Placebo laser therapy: patients receive the same treatment on the same area as experimental group for the same period without turning on the device.
  all 20 will receive Placebo laser therapy: patients receive the same treatment on the same area as experimental group for the same period without turning on the device.
  Interventions: Procedure: neural mobilization; Other: placebo laser therapy

INTERVENTIONS:
Device: Low Level Laser Therapy by (Eme Physio, Lasermed 2200), GaAs laser, 1 cm2 beam area,7,000 Hz, 17 mW, 1 J/cm2, Pesaro, Italy) — (Eme Physio, Lasermed 2200), GaAs laser, 1 cm2 beam area,7,000 Hz, 17 mW, 1 J/cm2, Pesaro, Italy) .
  Patient lies in side lying on the non-affected side which is opposite to the side of radicular pain, hip and knee in flexion 90. Twenty points were established for treatment, 12 over the lumbar spine, at the same Side of the radicular pain, from l2 to s1 vertebra, distance between these points is 2 cm. In the thigh, eight points were marked at equal distances from each other, four in the path of l5 root and four in the path of s1 root from hip to knee. The leaser probe is held in 90 degree over the skin with complete skin contact
  Arms: Experimental group (B)
Procedure: neural mobilization — Mobilization will be through using slump sitting maneuver (Both techniques slider and tensioner.
  •The slider neurodynamic mobilization technique: The patient moves actively and conversely from a position of neck and trunk flexion, knee flexion, and ankle plantar flexion, to a position of neck and trunk extension, knee extension and ankle dorsiflexion
  The tension neurodynamic mobilization technique:
  The patient moves actively and conversely from a position of neck and trunk extension, knee flexion, and ankle plantar flexion, to a position of neck and trunk flexion, knee extension, and ankle dorsiflexion
Other: placebo laser therapy — patients receive the same treatment on the same area as experimental group for the same period without turning on the device.
  Arms: control group (A)

SUMMARY:
This study attempts to answer the following research question: what is the combined effect of low level laser therapy and neural mobilization on lumber disc prolapse in decreasing pain, improving functional disability, improving neural mobility and improve lumber flexion mobility?

DETAILED DESCRIPTION:
Lumbar disc prolapse is a movement of disc material out of the intervertebral disc space. Protruded nucleus comes in contact with the surrounding nerves, causing their compression that in turn results in severe radicular pain.

The purpose of this study is to assess the combined effect of low level laser therapy and neural mobilization on lumber disc prolapse, this assessment will be done through assessment of pain, functional disability, neural mobility and lumber flexion mobility.

Subjects and Methods : 40 Patients with lumber disc prolapse and radiculopathy based on clinical examination by orthopedic surgeon and (MRI) imaging aged between 30 and 50 years . This study will be a double blinded randomized controlled trial .

After including patients in the study, they will be randomly assigned into 2groups :

Control group (A) (n=20): will receive placebo laser therapy plus neural mobilization.

Experimental group (B) (n=20): patients will receive low level laser therapy plus neural mobilization Both control group and experimental group receive infrared as warming up before treatment for12 sessions, each for 15 min, 3 days per week, for a period of 4 weeks .

All patients will perform all assessment procedures accurately (straight leg raising test, slump test and Schober's test ) and will fill (VAS) and (ODI) accurately.

Mobilization will be through using slump sitting maneuver (Both techniques slider and tensioner).Neural mobilization will be applied in form of 3 sets every set 10 repetitions and the end Position was hold for 5 seconds and the rest between sets was 5 minutes. All the patients will receive 12 sessions (3 times/week for 4 weeks).

: patients receive LLLT will lie in side lying on the non-affected side which is opposite to the side of radicular pain, hip and knee in flexion 90.Twenty points were established for treatment, 12 over the lumbar spine, at the same Side of the radicular pain and 8 points over thigh for 3 sessions per weak for 4 Weeks.

The hypotheses for this study are:

1. There will be significant improvement in pain after combination of LLLT and neural mobilization.
2. There will be significant improvement in functional disability after combination of LLLT and neural mobilization.
3. There will be significant improvement in lumber flexion mobility after combination of LLLT and neural mobilization.
4. There will be significant improvement in neural mobility after combination of LLLT and neural mobilization.

ELIGIBILITY:
Inclusion Criteria:

* 1-patients referred from orthopedic surgeon with diagnosis of lumbar disc prolapse and radiculopathy (subacute >3 weeks or chronic > 3 months and lasting up to 12 months) .

  2-Participants had MRI examination, which confirmed the diagnosis of lumber disc prolapse in addition of radiological changes in the intervertebral discs of the spine and affection of peripheral nerve root.

  3-Aged between 30 and 50 years .

Exclusion Criteria:

* 1- Patients who had undergone any surgical intervention in the spine. 2- Any other dysfunctions of the spine rather than lumber disc prolapse (fractures, tumors, spondylolisthesis, rheumatic diseases, and cauda equina syndrome).

  3- The patient is under any medical treatment. 4- Pregnancy, cardiovascular failure, pacemaker, metal implants, skin lesions in the treatment area.

  5- Neurological deficits such as myelopathy, lumber canal stenosis and Piriformis syndrome 6- Malignancy, systemic inflammatory disease, or infectious disease. 7- Acute lumber disc prolapse will be excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
pain assessment before and after treatment | 4 weeks
  by visual analog scale (VAS)
Functional disability :evaluate the patient's ability to perform various activities of daily living | 4 weeks
  by Oswestry Disability Index (ODI)
evaluate neural mobility before and after treatment | 4weeks
  by Straight leg raising test (SLR) ,The range of motion of the SLR test was measured as the angle of hip flexion in relation to the horizontal
evaluate lumbar flexion mobility before and after treatment | 4weeks
  by Schober's test
Neurological assessment screening of neuropathic pain | 4 weeks
  by slump test

CONTACTS AND LOCATIONS:
Overall Officials: Nasr A Abdelkader, PHD, Principal Investigator — Assistant professor, Department of physical therapy for musculoskeletal disorders and its surgeries
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No